CLINICAL TRIAL: NCT07029672
Title: Acute Respiratory Infections and Chronic Respiratory Disease Exacerbation Characterisation and Personalised Treatment Platform Study 2
Brief Title: The AcCREDiT 2 Study
Acronym: ACCREDIT2
Status: Not yet recruiting | Type: Observational
Sponsor: Manchester University NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: B02407
Record Dates: First submitted 2025-05-01; First posted 2025-06-19 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Chronic Respiratory Conditions; COPD; Pneumonia; Bacterial Infections; Viral Infections; Respiratory Exacerbation
Keywords: ACCREDIT
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Pneumonia; Bacterial Infections; Virus Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The ACCREDIT study - Acute respiratory infections and chronic respiratory disease exacerbations characterisation and personalised treatment platform study 2 (AcCREDiT 2).

Patients with respiratory infections (such as pneumonia) or exacerbations of chronic respiratory conditions (such as emphysema) often require hospital admission. Infections or exacerbation are commonly caused by bacteria, viruses or fungi. In at least a quarter of patients no infectious cause of the exacerbation is found. Depending on the cause of the respiratory infections or exacerbations of chronic respiratory condition patients require prompt treatment with anti-infective drugs (antibiotics, anti-fungal or antiviral drugs) or anti-inflammatory drugs such as corticosteroids.

Patients with respiratory infection or exacerbations of chronic respiratory conditions develop symptoms such as cough, sometimes with sputum, fever or breathlessness. These symptoms can be similar across several conditions, many of which are not due to infection (for example heart failure or blood clots in the lungs). When assessing patients with respiratory symptoms, clinicians face the challenge of limited information in the early stages of care as it takes three days to identify infectious organisms in the laboratory. Even when an infection is strongly suspected, distinguishing bacterial from viral or fungal infections on clinical grounds alone is difficult. This uncertainty often leads clinicians to prescribe a number of treatments, including antibiotics, before a clear diagnosis is made. Timely treatment is crucial for success and improved patient outcomes, especially for critically ill patients admitted to the intensive care unit (ICU). However, antibiotics may cause side effects, such as sickness and diarrhoea, and overuse of antibiotics leads to antibiotic resistance, making antibiotics less effective when they are really needed. Giving antibiotics to patients with an infection or exacerbation and avoiding antibiotics in patients without an infection requires rapid diagnostic tests. Furthermore, giving antibiotics prior to taking samples to diagnose infection can affect the sample being tested making it more likely to not give a useful result. For a diagnostic test for infection to be most useful it needs to be collected before an antibiotic is given - this is true for both clinical tests and those research tests which are clinical tests in development.

Modern technologies allow testing for an infection in hours rather than days. In order to understand how effective these technologies are, samples need to be taken from patients before they start treatment. In routine NHS care samples to test for infection should be taken before treatment has been started. However, in research studies samples are often taken up to a day after treatment has started which affects how effective the test is at finding infection. The forerunner to this study, called AcCREDiT, proposed investigating very rapid ways of identifying individuals with respiratory infection and exacerbation. However, the study team encountered challenges during the informed consent process, particularly with acutely unwell patients. Therefore, the AcCREDiT-2 was designed in collaboration with patients and public contributors to look at the feasibility of a modified informed consent process: verbal consent, assent for individuals with capacity to consent for themselves, and deferred consent.

AcCREDiT-2 will be an observational study, meaning that no treatment will be changed, and no experimental drugs or tests used to influence the clinical care of participants. AcCREDiT-2 will also be a 'feasibility study', which is a smaller study designed to see what works well before embarking on a larger project. During the study the investigators will collect clinical information and samples, such as blood, sputum and stool, from patients who come to hospital with a presumed respiratory infection or exacerbation of their chronic respiratory condition. The investigators will compare new diagnostic tests to traditional laboratory tests to understand their relative advantages and disadvantages for patient care.

This is a 'feasibility' study, a small study ran first to make sure things work properly before expanding to a much larger study.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Clinically suspected acute respiratory infection or exacerbation of chronic respiratory disease
* Availability of respiratory tract sample

  1. Spontaneously breathing patients are able to produce a sputum sample
  2. Mechanically ventilated patients in intensive care are due to have an Bronchoalveolar lavage or non-directed bronchial lavage for a clinical indication
* Due to receive either:

  1. an anti-infective agent (e.g. antibiotic, antiviral or antifungal) OR
  2. a systemic anti-inflammatory agent (e.g. corticosteroid)
* Valid informed consent, assent or enrolment through deferred consent
* Re-enrolment will be allowed if presenting for a separate acute event

Exclusion Criteria:

* Alternate respiratory cause of presentation in the opinion of the treating physician (e.g. pulmonary embolism, heart failure, etc.)
* High clinical likelihood of infection with a Hazard Group 3 pathogen (e.g. tuberculosis, anthrax, plague)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In patients whose symptoms are consistent with an acute respiratory infection or exacerbation, but the prescription of an eligible agent has not yet been confirmed
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Feasibility of timely recruitment, assessment, and retention during follow up | 12 months
  Endpoints: Number of patients recruited within 12 months of study start, recruitment expected at a minimum of 2 patients per week enrolled into the study, feasibility attainment target: 120 patients across different clinical environments and diagnostic categories.

SECONDARY OUTCOMES:
Efficacy of verbal consent | 12 months
  Feasibility of study - Proportion of patients declining consent at verbal consent stage
Efficacy of 'consent to continue' model following verbal consent | 12 months
  Measure of study feasibility - Proportion of patients voluntarily withdrawing from study following verbal consent
Availability of respiratory tract samples and stool samples for analysis | 12 months
  Measure of study feasibility - Proportion of patients in whom sputum and/or stool samples are successfully obtained for analysis
Infectious aetiology of presentation | 12 months
  Measure of study feasibility - Proportion of patients presenting with bacterial infection, viral infection, fungal infection, or no identifiable infective causes
Diagnostic categorisation of patients recruited | 12 months
  Study feasibility assessment - Proportion of patients presenting with prespecified diagnoses (e.g. pneumonia, exacerbation of COPD)
Performance of different diagnostic strategies | 12 months
  Measure of study feasibility - Comparison of results from routine microbiological approaches (service standard) with molecular techniques to identify pathogens.
Impact of delayed sampling on diagnosis and prescribing of antibiotics | 12 months
  Comparison of results from blood and sputum samples taken prior to treatment being commenced with samples collected 3-6 hours after treatment has been commenced.
Hospital length of stay (days) | 12 months
  Number of days from hospital admission to discharge - informing feasibility of study and future study
ICU length of stay, if admitted (days) | 12 months
  Number of days from ICU admission to discharge to inform feasibility of future study and recruitment methods
28-day mortality | 12 months
  Proportion of patients alive at 28 days from enrolment - feasibility of study and recruitment methods

CONTACTS AND LOCATIONS:
Locations (1):
- Manchester University NHS Foundation Trust, Manchester, United Kingdom